CLINICAL TRIAL: NCT04821960
Title: Improving Emotional Well-being and Quality of Life in Older Adults Experiencing Dementia-related Fear.
Brief Title: Memory and Fear Study (Fear of Memory Loss Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00214078
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Anxiety and Fear
Keywords: Mindfulness; Fear of memory loss
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Mindfulness Program (Active Comparator): Routine mindfulness lessons and activities.
  Interventions: Behavioral: Conventional Mindfulness Program
- Tailored Mindfulness Program for Fear of Memory Loss (Experimental): Tailored mindfulness lessons and activities for fear of memory loss.
  Interventions: Behavioral: Tailored Mindfulness Program for Fear of Memory Loss

INTERVENTIONS:
Behavioral: Tailored Mindfulness Program for Fear of Memory Loss — The tailored mindfulness program has been specifically created to focus on fear of memory loss compared to general mindfulness lessons and activities.
  Other Names: Conventional Mindfulness Program
  Arms: Tailored Mindfulness Program for Fear of Memory Loss
Behavioral: Conventional Mindfulness Program — Routine non-tailored mindfulness lessons and activities.
  Arms: Conventional Mindfulness Program

SUMMARY:
This study is a randomized control study to determine the impact of a tailored, web-based mindfulness program to reduce anxiety and increase the quality of life in older adults experiencing dementia-related fears, relative to a conventional meditation program.

DETAILED DESCRIPTION:
The study will test two different types of online mindfulness programs to see if an online self-paced mindfulness program can help reduce anxiety related to memory loss. Participants will be involved in the study for a total of 10 weeks. Participants will log on to an online mindfulness program 4 days per week for about 10-20 minutes each. The total program will last 3 weeks. Participants will also be asked to complete questionnaires before starting the program, during the program, and after they complete the program.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Elevated dementia-related fear
* Able to read/write in English
* Willingness to be randomized to intervention group
* Willingness to complete three weeks of self-guided intervention, questionnaires, and cognitive tests.
* Access to a reliable internet connection

Exclusion Criteria:

* Diagnosis of mild cognitive impairment, Alzheimer's Disease, or dementia by a healthcare provider.
* Impaired cognitive or neurologic function
* Unstable medical condition
* Severe depression
* Current treatment for anxiety or depression
* Current participation in another psychotherapy
* Current use of psychiatric medication
* Current substance use disorder
* Inadequate vision or hearing to interact with study materials

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared with other researchers.

REFERENCES:
- [Derived] Farina FR, Regan J, Marquez M, An H, O'Loughlin P, Pavithra P, Taddeo M, Knight RC, Bennett M, Lenaert B, Griffith JW. Reducing fear and avoidance of memory loss improves mood and social engagement in community-based older adults: a randomized trial. BMC Geriatr. 2023 Nov 29;23(1):786. doi: 10.1186/s12877-023-04470-4. PMID 38030988
- [Derived] O'Loughlin P, Pavithra P, Regan J, Bennett M, Knight R, Lenaert B, Marquez M, Taddeo M, Griffith J, Shapiro R, Farina F. A Randomized Controlled Trial Investigating the Feasibility of a Low-Intensity Psychological Intervention for Fear of Memory Loss and Quality of Life in Older Adults: Protocol for the Reducing Fear and Avoidance of Memory Loss (REFRAME) Study. JMIR Res Protoc. 2021 Jul 30;10(7):e30514. doi: 10.2196/30514. PMID 34328428

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Mindfulness Program | Tailored Mindfulness Program for Fear of Memory Loss
Started | 41 | 40
Completed | 36 | 30
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Mindfulness Program | Tailored Mindfulness Program for Fear of Memory Loss | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 28 | 48
  >=65 years | 21 | 12 | 33
Age, Continuous [Mean (Full Range); unit: years] | 63.7 [55.5 to 83.9] | 67 [55.1 to 90.2] | 65.4 [55.1 to 90.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 41 | 39 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 39 | 32 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 10 | 81

OUTCOME MEASURES:

1. Primary Outcome: Fear and Avoidance of Memory Loss (FAM) Scale Score at Follow-up
Description: A 24-item scale to assess fear of memory loss. Scores range from 24-120 points with a higher score indicating a higher fear of memory loss.
Time Frame: 10 Weeks Post-Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Mindfulness Program | Tailored Mindfulness Program for Fear of Memory Loss
Number analyzed (Participants) | 33 | 25
score on a scale | 63.9 (11.3) | 60.3 (10.6)

2. Primary Outcome: Fear of Alzheimer's Disease Scale (FADS) Score at Follow-up
Description: A 30-item scale to assess fear of Alzheimer's disease. Minimum score = 0; maximum score = 120. A higher score indicates a greater fear of developing Alzheimer's Disease.
Time Frame: 10 Weeks Post-Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Mindfulness Program | Tailored Mindfulness Program for Fear of Memory Loss
Number analyzed (Participants) | 40 | 33
score on a scale | 47.3 (20.7) | 45.2 (20)

3. Secondary Outcome: Memory Failure Scale (MFS)
Description: A 12-item scale that measures memory failure that people tend to experience in everyday life. Minimum score=12; maximum score= 60. A higher score indicates a greater likelihood of memory failures.
Time Frame: 10 Week Post-Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Mindfulness Program | Tailored Mindfulness Program for Fear of Memory Loss
Number analyzed (Participants) | 40 | 33
score on a scale | 34.9 (7.7) | 32.2 (8.5)

ADVERSE EVENTS:
Time Frame: Data were collected over a 10 week period.
Arm/Group | Conventional Mindfulness Program | Tailored Mindfulness Program for Fear of Memory Loss
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04821960/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT04821960/SAP_002.pdf
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04821960/ICF_001.pdf